CLINICAL TRIAL: NCT05357976
Title: The Effects of Body Mass Index on Thoracic Paravertebral Block Analgesia Treatment in Patients Undergoing Thoracoscopic Surgery
Brief Title: The Effects of Body Mass Index on Thoracic Paravertebral Block Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Nilgün Zengin, Principal İnvestigator, Ankara City Hospital Bilkent
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E.Kurul-E1-22-2596
Record Dates: First submitted 2022-04-25; First posted 2022-05-03 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Pain, Postoperative; Acute Pain; Thoracic Paravertebral Block; Body Mass Index; Thoracic Surgery, Video-Assisted
MeSH Terms: conditions — Pain, Postoperative; Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with a BMI of 18-24.9 kg/m2 (Active Comparator): The needle will be advanced to the paravertebral area with an ultrasound-guided in-plane technique. 30 ml of 0.25% bupivacaine will be injected into this area.
  Interventions: Procedure: Thoracic Paravertebral Block
- Patients with a BMI of 25-29.9 kg/m2 (Active Comparator): The needle will be advanced to the paravertebral area with an ultrasound-guided in-plane technique. 30 ml of 0.25% bupivacaine will be injected into this area.
  Interventions: Procedure: Thoracic Paravertebral Block
- Patients with a BMI of 30-40 kg/m2 (Active Comparator): The needle will be advanced to the paravertebral area with an ultrasound-guided in-plane technique. 30 ml of 0.25% bupivacaine will be injected into this area.
  Interventions: Procedure: Thoracic Paravertebral Block

INTERVENTIONS:
Procedure: Thoracic Paravertebral Block — Thoracic paravertebral block will be applied to the patients under real-time ultrasound guidance.

SUMMARY:
Obesity has become one of the world's leading health problems. It is known that obesity causes many diseases and negatively affects the quality of life. For this reason, many conditions that are thought to be effective in obesity and concern the quality of life of patients have been scientifically researched and continue to be investigated. One of them is postoperative pain. Although there are studies stating that there is no relationship between body mass index (BMI) and postoperative pain, when the literature data is examined, it is thought that obesity is a risk factor for postoperative pain and changes pain sensitivity and analgesic needs of patients. There are also studies in the literature stating that the level of postoperative pain increases in parallel with each unit increase in BMI.

After thoracic surgery, many analgesic methods have been suggested, including thoracic epidural analgesia (TEA), thoracic paravertebral block (TPVB), intercostal nerve blocks (ICSB), erector spina plane block (ESPB), serratus anterior plane block (SAPB). This study will compare the effects of BMI on postoperative pain in patients undergoing TPVB for postoperative analgesia and thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old
* ASA physical status I-II-III
* BMI 18 to 40 kg/m2
* Elective video-assisted thoracoscopic surgery

Exclusion Criteria:

* Patient refusing the procedure
* Emergency surgery
* Chronic opioid or analgesic use
* Patients who will operate under emergency conditions
* Patients who will not undergo VATS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-04-25 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-13 (Actual)

PRIMARY OUTCOMES:
Pain Scores | 1st hour after surgery.
  Pain will be assessed at the first-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Pain assessment will be done at the 1st, 2nd, 4th, 12th, 24th, and 48th hours after surgery.
Pain Scores | 2nd-hour after surgery.
  Pain will be assessed at the 2nd-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 4th-hour after surgery.
  Pain will be assessed at the 4th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 12th-hour after surgery.
  Pain will be assessed at the 12th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 24th-hour after surgery.
  Pain will be assessed at the 24th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 48th-hour after surgery.
  Pain will be assessed at the 48th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
Morphine Consumption | 24 hours after surgery
  Morphine consumption for 24 hours will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Nilgün Zengin, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara City Hospital, Çankaya, Ankara
  - Ankara Atatürk Chest Diseases and Thoracic Surgery Training and Research Hospital, Keçiören, Ankara

REFERENCES:
- [Derived] Zengin EN, Alagoz A, Yigit H, Sazak H, Sekerci S, Zengin M. The effect of body mass index on thoracic paravertebral block analgesia after video-assisted thoracoscopic surgery; a prospective interventional study. BMC Anesthesiol. 2023 Sep 4;23(1):297. doi: 10.1186/s12871-023-02264-0. PMID 37667207